CLINICAL TRIAL: NCT02817620
Title: Pilot Study to Assess Antioxidant Efficacy of a Spirulina Water Extract on Oxidized LDL Status and Lipids Metabolism on Subjects With Metabolic Syndrome
Brief Title: Study to Assess Antioxidant Efficacy of Spirulina on oxLDL and Lipids Metabolism on Subjects With Metabolic Syndrome
Acronym: SPIROX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Algosource (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC15039
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirulysat® (Experimental): Food supplement packaged in 10 ml vials called Spirulysat®. This product is a phycocyanin concentrated fresh spirulina water extract (Spirulina Platensis). 2 vials daily to consume in the morning, just before the breakfast, in a glass of water, during 12 weeks (from V1 to V3 visit).
  Interventions: Dietary Supplement: Spirulysat®
- Placebo (Placebo Comparator): Placebo with the same characteristics, appearance, packaging and composition as the active formula except for active ingredient (Spirulina) replaced by a classical blue food colorant used to colour desserts. 2 vials daily to consume in the morning, just before the breakfast, in a glass of water, during 12 weeks (from V1 to V3 visit).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Spirulysat®
  Arms: Spirulysat®
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to assess the beneficial effect of a spirulina water extract (product named Spirulysat®) compared to a placebo in the blood level ratio of oxidized LDL / total LDL cholesterol in subjects with metabolic syndrome after 12 weeks of consumption

ELIGIBILITY:
Inclusion Criteria:

To be eligible to the study, male and female volunteers will have to fulfil the following criteria (assessment based on the medical examination performed at V0 with a checking at V1):

* Age between 18 and 65 years (limits included),
* BMI between 25 and 35 kg/m² (limits included),
* With metabolic syndrome defined as central obesity : waist circumference > 94 cm for man and > 80 cm for woman associated to at least 2 observed criteria among : Fasting blood triglycerides > 1.5 g/L and/or Fasting blood HDL cholesterol < 0.4 g/L for man and < 0.5 g/L for woman and/or Fasting blood glucose level > 1 g/L and/or Arterial pressure > 130/85 mmHg or under antihypertensive treatment,
* For women : non menopausal with the same reliable contraception since at least 3 months before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicide gel accepted) or menopausal without or with hormone replacement therapy started at stable dose since at least 3 months before the beginning of the study and agreeing to keep it during the entire duration of the study,
* Weight stable with +/- 5 % in the last 3 months ,
* Non smoking or with tobacco consumption < 10 cigarettes / day,
* Good general and mental health with in the opinion of the investigator : no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agree to be registered on the volunteers in biomedical research file,

After V0 biological analysis the subjects will be eligible to the study on the following criterion :

* Blood fasting lipid profile not requiring therapeutic intervention meaning professional recommendations (AFSSAPS, 2005).

A re-screening can occur from 2 months after the exit of the study for failure to comply with one or more of the inclusion criteria listed above.

Exclusion Criteria:

Volunteers with the following criteria will be considered as non eligible to the study (assessment based on the medical examination performed at V0 with a checking at V1):

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble...,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* With a history of ischemic cardiovascular event,
* Having undergone recent surgical procedure (less than 6 months),
* Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg),
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient,
* Pregnant or lactating women or intending to become pregnant within 4 months ahead,
* Under cholesterol and/or lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 3 months before the V0 visit,
* Under medication which could affect blood lipid parameters (e.g. long-term corticosteroid systemic drug, systemic antibodies, androgens or enzyme inducers, etc.) or stopped less than 3 months before the V0 visit (antihypertensive stable long-term treatment tolerated),
* Regular intake of dietary supplements or "functional foods" which are known to have an impact on lipid metabolism (e.g. rich in plant stanol or sterol like PRO-ACTIV or DANACOL products, red yeast rice, policosanol, capsules containing omega-3 fatty acids from fish oils, etc.) or stopped less than 3 months before the V0 visit,
* Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the V0 visit,
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study,
* With a current or planned in the next 4 months specific diet (hyper or hypocaloric, vegan, vegetarian...) or stopped less than 3 months before the V0 visit,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Who made a blood donation in the 3 months before the V0 visit or intending to make it within 4 months ahead,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency,

After V0 biological analysis the subjects will be considered as non eligible to the study on the following criteria :

* Fasting blood triglycerides > 3.5 g/L (3.95 mmol/L),
* Blood ASAT, ALAT or GGT (Gamma Glutamyl Transferase) > 3xULN (Upper Limit of Normal),
* Blood urea > 12.11 mmol/L (value corresponding to 1.5xULN) or creatinine > 125 µmol/L,
* Blood hsCRP > 10 mg/L,
* Complete blood count with clinically significant abnormality according to the investigator.

A re-screening can occur from 2 months after the exit of the study for failure to comply with one or more of the exclusion criteria listed above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Changes in the ratio of fasting blood concentrations oxidized LDL / total LDL cholesterol | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in mU/g

SECONDARY OUTCOMES:
Changes in the ratio of fasting blood concentrations oxidized LDL / total LDL cholesterol | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in mU/g
Changes in fasting blood oxidized LDL level | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in mU/L
Changes in fasting blood oxidized LDL level | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in mU/L
Changes in fasting blood concentrations of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of hsCRP | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in mg/L
Changes in fasting blood concentrations of hsCRP | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in mg/L
Changes in fasting blood concentration of total free fatty acid | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in mmol/L
Changes in fasting blood concentration of total free fatty acid | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in mmol/L
Changes in fasting blood concentration of alkaline phosphatase | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentration of alkaline phosphatase | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentrations of ASAT (Aspartate aminotransferase) and ALAT (alanine aminotransferase) | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentrations of ASAT (Aspartate aminotransferase) and ALAT (alanine aminotransferase) | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentration of total antioxidant status | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in mmol/L
Changes in fasting blood concentration of total antioxidant status | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in mmol/L
Changes in concentration of urinary isoprostane (F2-isoprostane alpha) | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in ng/mL
Changes in concentration of urinary isoprostane (F2-isoprostane alpha) | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in ng/mL

OTHER OUTCOMES:
Bile acids levels in stool (desoxycholic acid, lithocholic acid, cholic acid, chenodesoxycholic acid, bile salt, ursodesoxycholic acid) | Baseline
Bile acids levels in stool (desoxycholic acid, lithocholic acid, cholic acid, chenodesoxycholic acid, bile salt, ursodesoxycholic acid) | 6 weeks
Bile acids levels in stool (desoxycholic acid, lithocholic acid, cholic acid, chenodesoxycholic acid, bile salt, ursodesoxycholic acid) | 12 weeks
Short chain fatty acids levels in stool (acetic acid, n-butyric acid, iso-butyric acid, n-valerianic acid, propionic acid) | Baseline
Short chain fatty acids levels in stool (acetic acid, n-butyric acid, iso-butyric acid, n-valerianic acid, propionic acid) | 6 weeks
Short chain fatty acids levels in stool (acetic acid, n-butyric acid, iso-butyric acid, n-valerianic acid, propionic acid) | 12 weeks
Blood level of Glutathione peroxidase | Baseline
Blood level of Glutathione peroxidase | 6 weeks
Blood level of Glutathione peroxidase | 12 weeks
Superoxide dismutase blood level | Baseline
Superoxide dismutase blood level | 6 weeks
Superoxide dismutase blood level | 12 weeks
Catalase blood level | Baseline
Catalase blood level | 6 weeks
Catalase blood level | 12 weeks
Intestinal microbiota (bacterial DNA extraction in stool) | Baseline
Intestinal microbiota (bacterial DNA extraction in stool) | 12 weeks
PON-1 (paraoxonase-1) in blood (arylesterase activity) | Baseline
PON-1 (paraoxonase-1) in blood (arylesterase activity) | 12 weeks
Body weight | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in kg
Body weight | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in kg
Total energy intake | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in kcal/day
Total energy intake | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in kcal/day
Percentage of energy intake from fat | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in %
Percentage of energy intake from fat | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in %
Percentage of energy intake from carbohydrates | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in %
Percentage of energy intake from carbohydrates | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in %
Percentage of energy intake from protein | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in %
Percentage of energy intake from protein | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in %
Dietary fiber intake | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in g/day (absolute quantities)
Dietary fiber intake | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in g/day (absolute quantities)
Saturated fatty acid intake | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in g/day (absolute quantities)
Saturated fatty acid intake | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in g/day (absolute quantities)
Mono-unsaturated fatty acid intake | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in g/day (absolute quantities)
Mono-unsaturated fatty acid intake | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in g/day (absolute quantities)
Poly-unsaturated fatty acid intake | 6 weeks
  Defined as the difference V2 (6 weeks) - V1 (baseline) in g/day (absolute quantities)
Poly-unsaturated fatty acid intake | 12 weeks
  Defined as the difference V3 (12 weeks) - V1 (baseline) in g/day (absolute quantities)
Heart rate (bpm) | Pre-inclusion (V0), Baseline (V1), 6 weeks (V2) and 12 weeks (V3)
Systolic blood pressure (mmHg) | Pre-inclusion (V0), Baseline (V1), 6 weeks (V2) and 12 weeks (V3)
Diastolic blood pressure (mmHg) | Pre-inclusion (V0), Baseline (V1), 6 weeks (V2) and 12 weeks (V3)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SCHMID, Study Director — Biofortis Mérieux NutriSciences; David GENDRE, Principal Investigator — Biofortis Mérieux NutriSciences
Locations (1):
- Biofortis Mérieux NutriSciences Clinical Investigation Center, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: Undecided